CLINICAL TRIAL: NCT04286347
Title: Pre-Surgery Assessing HCV, HBV, HIV Status and Revealing During Consultation With Anesthesiologist
Brief Title: HCV, HBV, HIV Testing During Consultation With Anesthesiologist
Acronym: SAHARA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding to continue any longer
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP191114; 2019-A03071-56 (Other: RCB)
Record Dates: First submitted 2020-01-17; First posted 2020-02-27 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: HCV; HBV; Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — HIV Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HCV, HBV, HIV testing (Experimental): All patient ≥ 18 years-old with a next planned surgery in Lariboisiere Hospital, Paris, France, able to give written informed consent for testing will be proposed to be tested for HIV and HCV if no previous testing found in the medical record and will be proposed to be tested for HBV if the patient belong to a high-risk group: high prevalence area (Asia, sub-Saharan Africa, French Indies, East and South Europe, North-Africa, Middle-East, India, Pakistan, South-America), IVDU, prisoners, unprotected sexual intercourses.
  Interventions: Procedure: HCV, HBV, HIV tests

INTERVENTIONS:
Procedure: HCV, HBV, HIV tests — HCV, HBV, HIV testing during consultation with Anesthesiologist before a planned surgery

SUMMARY:
The aim of the study is to assess the feasibility of HCV, HBV, HIV testing (according to the national guidelines) during consultation with Anesthesiologist before a planned surgery in Lariboisiere Hospital, Paris, France. The feasibility will be the number of tested patients divided by the number of patients who should have been tested according to the national guidelines (for each virus).

DETAILED DESCRIPTION:
The aim of the study is to assess the feasibility of HCV, HBV, HIV testing during consultation with Anesthesiologist before a planned surgery in Lariboisiere Hospital, Paris, France.

The national guidelines recommend at least one HIV testing during life and, more recently, one HCV testing during life to eradicate HCV infection. HBV testing is recommended in patients coming from high prevalence countries, IVDU, prisoners, patients with multiple sexual partners.

The feasibility will be the number of tested patients divided by the number of patients who should have been tested according to the national guidelines (for each virus).

HIV testing will use finger-stick whole blood (FSB) INSTI® HIV-1 & HIV-2 Rapid Antibody Test FSB (BioLytical TM Laboratories Inc., Richmond, B.C., Canada), with a sensitivity 99% [96.3-99.7] and a specificity 99.3%.

HCV testing will use finger-stick whole blood (FSB) Oraquick® HCV test, with a sensitivity and a specificity 99.1 and 100% respectively.

HBV testing will use finger-stick whole blood (FSB) Vikia® HBs Ag test, bioMérieux with a sensitivity and a specificity 96.5 and 99.9% respectively.

ELIGIBILITY:
Inclusion Criteria:

* patient ≥ 18 years-old
* planned surgery in Lariboisiere Hospital, Paris, France
* able to give written informed consent for testing
* proposed to be tested for HIV and HCV if no previous testing found in the medical record
* proposed to be tested for HBV if the patient belong to a high-risk group: high prevalence area (Asia, sub-Saharan Africa, French Indies, East and South Europe, North-Africa, Middle-East, India, Pakistan, South-America), IVDU, prisoners, unprotected sexual intercourses.

Exclusion Criteria:

* patient < 18 years-old
* emergency surgery
* unable to give written informed consent for testing: psychiatric diseases, neurologic diseases, …
* a previous testing for HIV and HCV found in the medical record and no obvious risk factor after previous testing
* the patient does not belong to a high-risk group for HBV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Feasibility of HCV, HBV, HIV testing | Day 0 : during initial consultation, up to 1 hour
  Feasibility (assessed by the number of tested patients divided by the number of patients who should have been tested according to the national guidelines (for each virus)) of HCV, HBV, HIV testing during consultation with Anesthesiologist before a planned surgery in Lariboisiere Hospital, Paris, France

SECONDARY OUTCOMES:
Acceptability of HCV, HBV, HIV testing | Day 0 : during initial consultation, up to 1 hour
  Acceptability (number of patients who accept to be tested divided by the number of patients who should have been tested according to the national guidelines (for each virus) of HCV, HBV, HIV testing during consultation with Anesthesiologist before a planned surgery in Lariboisiere Hospital, Paris, France
Acceptability of being treated (for each virus) for the patients who have been tested positive for HCV and/or HBV and/or HIV, by questionning | during Day 0, after the initial consultation
  Acceptability of being treated (for each virus) for the patients who have been tested positive for HCV and/or HBV and/or HIV during consultation, by direct questionning, with Anesthesiologist before a planned surgery in Lariboisiere Hospital, Paris, France.

CONTACTS AND LOCATIONS:
Locations (1):
- Lariboisière, Paris, France

IPD SHARING:
Plan to Share IPD: No